CLINICAL TRIAL: NCT04517357
Title: A Phase 2 Open Label, Randomised, Controlled, Multi-centre Study to Assess the Efficacy and Safety of Fluzoparib Combined With Apatinib Versus Fluzoparib Monotherapy in the Treatment of Relapsed Ovarian Cancer Patients
Brief Title: A Phase 2 Trial of Fluzoparib Combined With Apatinib Versus Fluzoparib Monotherapy in Treatment With Relapsed Ovarian Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-II-201
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Relapsed Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety Lead-in or Parallel， Fluzoparib+Apatinib (Experimental): Participants will receive Fluzoparib-Apatinib combination until progression
  Interventions: Drug: Fluzoparib+Apatinib
- Fluzoparib monotherapy (Active Comparator): Participants will receive Fluzoparib monotherapy until progression
  Interventions: Drug: Fluzoparib
- Exploratory cohort: Fluzoparib+Apatinib (Other): Participants who has previously received PARP inhibitor, will receive Fluzoparib-Apatinib combination until progression
  Interventions: Drug: Fluzoparib+Apatinib

INTERVENTIONS:
Drug: Fluzoparib+Apatinib — Fluzoparib-Apatinib combination
  Arms: Safety Lead-in or Parallel， Fluzoparib+Apatinib
Drug: Fluzoparib — Fluzoparib monotherapy
  Arms: Fluzoparib monotherapy
Drug: Fluzoparib+Apatinib — Fluzoparib-Apatinib combination
  Arms: Exploratory cohort: Fluzoparib+Apatinib

SUMMARY:
This is a multicenter, randomized, open-label, 2-arm Phase 2 study to evaluate the efficacy and safety of Fluzoparib with Apatinib versus Fluzoparib alone, as treatment, in relapsed ovarian cancer patients. The study contains a Safety Lead-in Phase in which the safety and tolerability of Fluzoparib+Apatinib will be assessed prior to the Phase 2 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed high-grade serous or endometrioid recurrent ovarian,fallopian tube,or peritoneal cancer.
2. Patients must have received at least 2 previous platinum-containing regimens.
3. At least one target lesion.
4. ECOG performance status 0-1.
5. Adequate bone marrow, kidney and liver function.

Exclusion Criteria:

1. Prior treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor or Apatinib.For exploratory cohort ，patients who received PARP inhibitor are eligible;
2. Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry. Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix allowed;
3. Radiation or anti-hormonal therapy or anticancer therapy within 14 days before first administration;
4. Known to be human immunodeficiency virus positive;
5. Known active hepatitis C virus, or known active hepatitis B virus;
6. Untreated and/or uncontrolled brain metastases;
7. Patients with clinical symptoms of cancer ascites, pleural effusion, who need to drainage, or who have undergone ascites drainage within 3 months prior to the first administration;
8. Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
(Safety Lead-in) dose limited toxicity (DLT) of Fluzoparib+Apatinib in the first cycle | up to 28 days
(Safety Lead-in) Recommended Phase II Dose (RP2D) of Fluzoparib+Apatinib | up to 28 days
(Phase 2) Objective response rate（ORR） in relapsed ovarian cancer patients | Assessed up to a maximum of 20 months
  Defined as Objective response rate per RECIST 1.1 criteria according to Investigator's assessment
(Exploratory research) Objective response rate（ORR） in relapsed ovarian cancer patients | Assessed up to a maximum of 20 months
  Defined as Objective response rate per RECIST 1.1 criteria according to Investigator's assessment

SECONDARY OUTCOMES:
AEs+SAEs | from the first drug administration to within 30 days for the last treatment dose
  Adverse Events and Serious Adverse Events
Progression free survival (PFS) | up to 20 months
  Defined as Progression free survival per RECIST 1.1 criteria according to Investigator's assessment
Disease control rate (DCR) | up to 20 months
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST 1.1
Duration of response (DoR) | up to 20 months
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response
Response rate by RECIST 1.1 criteria | up to 20 months
Response rate by GCIG CA125 | up to 20 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided